CLINICAL TRIAL: NCT04611477
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Efficacy of Synbiotic 365 on Body Composition in Overweight and Obese Individuals.
Brief Title: Effect of Synbiotic 365 on Body Composition in Overweight and Obese Individuals
Acronym: Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: NI/190701/SYNBIOTIC365/OO
Record Dates: First submitted 2020-09-28; First posted 2020-11-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2020-09

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): One capsule/day to be taken orally 30 minutes before breakfast
  Interventions: Other: Rice Hulk
- Synbiotic365 Ver 5 (Active Comparator): One capsule/day to be taken orally 30 minutes before breakfast
  Interventions: Other: Synbiotic365 Ver 5
- Synbiotic365 Ver 7 (Active Comparator): One capsule/day to be taken orally 30 minutes before breakfast
  Interventions: Other: Synbiotic365 Ver 7

INTERVENTIONS:
Other: Rice Hulk — Placebo
  Arms: Placebo
Other: Synbiotic365 Ver 5 — Active Comparator
  Arms: Synbiotic365 Ver 5
Other: Synbiotic365 Ver 7 — Active Comparator
  Arms: Synbiotic365 Ver 7

SUMMARY:
Evaluate the effect of Synbiotic 365 (Version 5 and 7) on body composition in overweight and obese individuals as measured by change in body mass index (BMI) and the percentage of body fat from Day 0 to Day 84 when compared to placebo by Dual Energy X-ray Absorptiometry scan (DEXA) for body composition (Body Mass Index, Lean Body Mass, Body Fat, Fat Free Mass).

ELIGIBILITY:
Participants meeting ALL of the following criteria will be recruited for the trial:

Inclusion:

1. Male and female participants aged ≥30 and ≤60 years.
2. Participants with a BMI in the range of ≥25 to 34.9 kg/m2.
3. Normal levels of SGOT and SGPT i.e. up to 2.5 times of upper limit of reference range.
4. Normal level of Creatinine i.e. up to 1.5 times of upper limit of reference range.

5 Alkaline Phosphatase i.e. up to 1.5 times of upper limit of reference range

6. Participants having At least 3 of the following five metabolic risk factors: i. Waist circumference: Men: ≥ 102 cm (40.15 inches); Women ≥88 cm (34.65 inches) ii. Triglycerides levels >150 mg/dL iii. Blood pressure ≥130 mm Hg (systolic, SBP) and/or ≥85 mm Hg(diastolic, DBP); iv. Fasting blood glucose ≥ 100 mg/ dL v. Low HDL level: Men: < 40 mg/dL; Women: < 50 mg/dL..

7. Participants willing to complete all the study procedures including study-related questionnaires and comply with the study requirements.

8. Participants willing to abstain from the restricted supplements and medications prior to inclusion and throughout the study period.

9. Participants ready to give voluntary, written, informed consent to participate in the study.

10. Participants willing to continue the same diet and exercise regime throughout the study period.

Exclusion:

1. Individuals having a history of smoking or currently smoking and also using any form of tobacco preparations.
2. Participants diagnosed with type II diabetes mellitus or undiagnosed cases of hyperglycemia with fasting blood sugar > 170 mg/dl.
3. Participants with blood pressure ≥150 mm Hg (systolic, SBP) and/or ≥ 99 mm Hg (diastolic, DBP)
4. Inability to walk independently
5. History of significant weight instability (defined as > 2 kg of weight loss over last 3 months)
6. Participants currently on diuretics, metformin or thyroid supplements. Presence of unstable, acutely symptomatic, or life-limiting illness.
7. Any significant neurological and psychiatric condition which may affect the participation and inference of the study's end points.

8 Unwillingness or inability to be randomized to any one of the three intervention groups.

9 Continuous participation in randomly assigned lifestyle intervention program for six months.

10 Bilateral hip replacements.

11 Unable to give consent.

12 Known cases of hypothyroidism.

13 Abnormal TSH value, out of reference range (<0.4μIU/mL and > 4.0μIU/mL).

14 Females with the history of irregular menses or any other gynecological disorder such as (polycystic ovarian syndrome (PCOS), hormonal disturbances, etc).

15 History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic disorders, that in the judgment of the investigator, would interfere with the participant's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the participant at undue risk.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2021-10-29 (Actual)

PRIMARY OUTCOMES:
Change in body mass index (BMI) and the percentage of body fat f | Day 0 (Baseline) to Day 84
  To investigate the effect of Synbiotic 365 (Version 5 and 7) on body composition in overweight and obese individuals as measured by change in body mass index (BMI) and the percentage of body fat from Day 0 to Day 84 when compared to placebo by Dual Energy X-ray Absorptiometry scan (DEXA) for body composition

SECONDARY OUTCOMES:
• Total body weight change in comparison to placebo on day 28, 56 and 84, from baseline, as assessed by weighing scale method. | Day 0 (Baseline) to Day 84
• Change in central obesity in comparison to placebo on day 28, 56 and 84, from baseline as assessed by the anthropometric index of waist-to-hip ratio. | Day 0 (Baseline) to Day 84
• Change in coronary risk in comparison to placebo on day 84 from baseline. | Day 0 (Baseline) to Day 84
• Change in blood glucose metabolism in comparison to placebo on day 84 from baseline as assessed by HOMA-IR [(fasting Glucose x fasting Insulin) /405)]. | Day 0 (Baseline) to Day 84
• Change in systemic inflammation in comparison to placebo on day 84 from baseline as assessed by hs-CRP test. | Day 0 (Baseline) to Day 84
• Change in health-related quality of life (HRQL) scores in comparison to placebo on day 28, 56 and 84 from baseline, as assessed by Gastrointestinal Quality of Life Index (GIQLI). | Day 0 (Baseline) to Day 84
• Change in satiety in comparison to placebo on day 28, 56 and 84, from baseline as assessed by the Three-Factor Eating Questionnaire (TFEQ) for satiety. | Day 0 (Baseline) to Day 84
• The change in vital signs monitoring on all the study visits from baseline. | Day 0 (Baseline) to Day 84
• The change in liver and renal safety parameters. | Day 0 (Baseline) to Day 84
• Adverse and serious adverse events recorded during the study duration on IP consumption, as compared to placebo. | Day 0 (Baseline) to Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Parag Dr. Salvi, MD, Principal Investigator — Shri Madhumadhav Clinic
Locations (1):
- Shri Madhumadhav Clinic, Mumbai, Maharashtra, India